CLINICAL TRIAL: NCT01771419
Title: Comparison Of Loop-Tip Wire Vs Tradictional Technique In The Cannulation Of The Common Bile Duct
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital San Paolo (Other)
Responsible Party: Principal Investigator, Benedetto Mangiavillano, MD, Hospital San Paolo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H San Paolo
Record Dates: First submitted 2013-01-15; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Post-ERCP Pancreatitis
Keywords: loop-tip; ERCP; cannulation of CBD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- loop-tip arm (Experimental): The cannulation of CBD will be obtained using the loop-tip wire (Cook Medical inc.)
  Interventions: Device: Loop-tip wire (Cook Medical) for the cannulation of the CBD
- Control arm (Active Comparator): The cannulation of CBD will be obtained with a Cook Medical sphincterotome CT-25 mm (tradictional technique)
  Interventions: Device: Cannulotome CT-25mm Cook Medical

INTERVENTIONS:
Device: Loop-tip wire (Cook Medical) for the cannulation of the CBD
  Arms: loop-tip arm
Device: Cannulotome CT-25mm Cook Medical
  Arms: Control arm

SUMMARY:
Selective cannulation of common bile duct (CBD) by insertion of a guide-wire seems to be associated with fewer complications and post-ERCP (Endoscopic retrograde cholangiopancreatography) pancreatitis (PEP) rate than the conventional biliary tree access with cannulotome (CT-25 Cook Medical) with contrast injection even if results are conflicting. the aim of our study is to test a new guide-wire (loop-tip wire), with a loop in the tip, for the prevention of PEP and biliary tree access, in PEP high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* high-risk patients for post-ERCP pancreatitis

Exclusion Criteria:

* age < 18 years
* allargy to the contrast medium
* previous biliary or gastric surgery
* neoplastic patients
* previous biliary or pancreatic sphincterotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-02 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
post ERCP pancreatitis rate | up to 4 weeks
  participants will be followed for the duration of hospital stay, an expected average of 2 weeks

SECONDARY OUTCOMES:
Number of attempts to obtain the cannulation of CBD and number of participants with adverse events as a measure of safety and tolerability | up to 4 weeks
  participants will be followed for the duration of hospital stay, an expected average of 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- San Paolo Hospital, Milan, Italy, Italy

REFERENCES:
- [Derived] Masci E, Mangiavillano B, Luigiano C, Bizzotto A, Limido E, Cantu P, Manes G, Viaggi P, Spinzi G, Radaelli F, Mariani A, Virgilio C, Alibrandi A, Testoni PA. Comparison between loop-tip guidewire-assisted and conventional endoscopic cannulation in high risk patients. Endosc Int Open. 2015 Oct;3(5):E464-70. doi: 10.1055/s-0034-1392879. Epub 2015 Sep 15. PMID 26528503